CLINICAL TRIAL: NCT05447195
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Efficacy and Safety of CAN008 Plus TMZ During and After Radiation Therapy in Subjects With Newly Diagnosed Glioblastoma
Brief Title: Phase 2 Study of CAN008 in Subjects With GBM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CANbridge Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN008-G-202; CTR20211888 (Registry Identifier: Center For Drug Evaluation, NMPA, China)
Record Dates: First submitted 2022-06-17; First posted 2022-07-07 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Newly-diagnosed Glioblastoma
Keywords: Glioblastoma; CAN008; APG101
MeSH Terms: conditions — Glioblastoma | interventions — APG101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blinded. Except for the non-blinded team, no other participants associated with this study should attempt to learn the treatment group assignment or which study treatment they are receiving.The unblinding of all subjects must be carried out after the database is locked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAN008 (Experimental): CAN008 IV infusion weekly
  Interventions: Drug: CAN008
- placebo (Placebo Comparator): Placebo IV infusion weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAN008 — Treatment in this study is divided into four periods. Period 1 (W1-W6) is the triple therapy period in which subjects in both groups will be given CAN008 + RT + TMZ. Period 2 (W7-W10) is the treatment-free (rest) period in which subjects do not receive any study drug/therapy. Period 3 (W11-W58) is the CAN008+TMZ maintenance therapy period in which subjects in both groups are given CAN008+TMZ. Period 4 (after W59) is the monotherapy period in which subjects are given CAN008 IV infusion weekly until disease progression.
  Other Names: APG101
  Arms: CAN008
Drug: Placebo — Treatment in this study is divided into four periods. Period 1 (W1-W6) is the triple therapy period in which subjects in both groups will be given placebo + RT + TMZ. Period 2 (W7-W10) is the treatment-free (rest) period in which subjects do not receive any study drug/therapy. Period 3 (W11-W58) is the placebo+TMZ maintenance therapy period in which subjects in both groups are given placebo+TMZ. Period 4 (after W59) is the monotherapy period in which subjects are given placebo IV infusion weekly until disease progression.
  Arms: placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled Phase 2 study whose objectives are to evaluate the clinical efficacy and safety of CAN008 plus TMZ during and after radiation therapy in newly-diagnosed subjects with glioblastoma who have undergone surgical excision.

DETAILED DESCRIPTION:
This study plans to enroll approximately 117 subjects. Subjects determined as having met inclusion criteria through screening will be randomized into treatment groups (CAN008 + RT + TMZ, 78 subjects) and the control group (placebo + RT + TMZ, 39 subjects) in a ratio of 2:1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70.
* Newly diagnosed glioblastoma.
* Tumor excision rate ≥80%.
* Karnofsky performance score ≥70.

Exclusion Criteria:

* Medical history of brain radiation therapy or electric field treatment of tumor.
* Primary infratentorial glioblastoma, multifocal glioma (≥ 2), or leptomeningeal metastasis.
* Any malignant tumor (excluding WHO grade I-II low-grade astrocytomas, basal cell carcinoma, and carcinoma in situ).
* Receiving high-dose hormone therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  To evaluate the efficacy of CAN008 plus temozolomide (TMZ) treatment in subjects with newly diagnosed glioblastoma (GBM) during and after radiation therapy

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China